CLINICAL TRIAL: NCT03757650
Title: THE EFFECT OF HELICOBACTER PYLORI ERADICATION THERAPY TO GASTRIC WALL THICKNESS BEFORE THE LAPAROSCOPIC SLEEVE GASTRECTOMY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ANIL ERGIN, Dr Anil ERGIN , General Surgery , Asistant doctor, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ANIL ERGIN
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Helicobacter Pylori Infection; Obesity, Morbid
Keywords: obesity; laparoscopic sleeve gastrectomy; helicobacter pylori; gastric wall thickness
MeSH Terms: conditions — Obesity, Morbid; Obesity | interventions — bismuth subsalicylate; Amoxicillin; Clarithromycin; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- HP eradication therapy positive-HP positive (Active Comparator): who has HP positive endoscopic biopsy will take HP eradication therapy one month before the surgery
  Interventions: Drug: Bismuth Subsalicylate
- HP eradication therapy negative-HP positive (Active Comparator): who has HP positive endoscopic biopsy and will not take any medication about HP
  Interventions: Drug: Bismuth Subsalicylate
- HP negative-Control group (No Intervention): who has HP negative endoscopic biopsy and will not take any medication. (control group)

INTERVENTIONS:
Drug: Bismuth Subsalicylate — omeprazole 2x1) + clarithromycin 2x500 mg + amoxicilline 2x1000 mg + Bismuth Subsalicylate 2x1
  Other Names: amoxicillin; clarithromycin; omeprazole
  Arms: HP eradication therapy negative-HP positive; HP eradication therapy positive-HP positive

SUMMARY:
Laparoscopic sleeve gastrectomy is one of the most popular bariatric surgery in the world. The most important complication about this surgery that the leakage from the stapler line because of the inconvenient stapler choice..The stapler colour has to be chosen to the gastric wall thickness. It is not known well that the effect of Helicobacter pylori to gastric wall thickness Nobody pay any attention about being Helicobacter pylori positive when they are choosing stapler colour during the Laparoscopic sleeve gastrectomy so that everybody use the same type of stapler in Helicobacter pylori positive and negative patients during the Laparoscopic sleeve gastrectomy .Because of this inconvenient staplers use in the Laparoscopic sleeve gastrectomy the risk of leakage would be increase. Purpose of this research is that what is the effect of Helicobacter pylori to the gastric wall thickness and if the patients who will undergo Laparoscopic sleeve gastrectomy take the Helicobacter pylori eradication therapy before the surgery will gastric wall thickness increase or decrease. .

DETAILED DESCRIPTION:
All patients who will undergo to Laparoscopic sleeve gastrectomy have upper gastrointestinal system endoscopy before the surgery in our clinical routine. In our research some patients who has Helicobacter pylori positive endoscopic biopsy will take Helicobacter pylori eradication therapy one month before the surgery and some patients will not take any medication about Helicobacter pylori. All of gastric specimens( Helicobacter pylori positive or negative ) will examine microscopically in the pathology laboratory. The two groups which preoperatively Helicobacter pylori positive detected in endoscopic biopsy will compare with Helicobacter pylori negative control group. Control group will include 30 patients. The other two groups will include 44 patients for each group . The number of patients of group has been determined by power analysis. Gastric specimen will be examined by 3 points ; fundus, corpus, antrum. All of microscopic measurements will be done from that points from minor curvatura. These 3 points ; fundus( 1 cm from the top of staple line) , corpus (middle of the staple line) , antrum ( 1 cm far from the bottom of staple line ). All these points 5 mm far from the minor curvatura. These 3 points will examine about wall thickness (mucosa- submucosa-muscularis propria -serosa ) and the status of Helicobacter pylori. The end of the study it can be determined the effect of Helicobacter pylori to the gastric wall thickness.

ELIGIBILITY:
Inclusion Criteria:

* All patients who will undergo to LSG will have upper gastrointestinal system endoscopy before the surgery and positive HP results.

Exclusion Criteria:

* Having allergy to the medications which use for the HP eradication therapy
* The patients who is incompatible for the HP eradication therapy
* The patients who decided to undergo to another bariatric surgery peroperatively

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
measurements of gastric wall thickness | one month
  The effect of Helicobacter Pylori eradication therapy to the gastric wall thickness

SECONDARY OUTCOMES:
Choosing the correct stapler colour during Laparoscopic Sleeve Gastrectomy by accounting gastric wall thickness thanks to knowing effect of HP positivity to gastric wall thickness | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Sultan Mehmet Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No